CLINICAL TRIAL: NCT07112053
Title: A Phase II Study of STEMVAC Vaccine Therapy for Patients With Hormone Receptor Positive Metastatic Breast Cancer
Brief Title: A Vaccine (STEMVAC) With Standard Endocrine-Based Therapy or Chemotherapy for the Treatment of Metastatic Hormone Receptor Positive, HER2 Negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG1125521; NCI-2025-04692 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0020922 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2025-07-18; First posted 2025-08-08 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic HER2-Negative Breast Carcinoma; Metastatic Hormone Receptor-Positive Breast Carcinoma
MeSH Terms: interventions — Capecitabine; Cyclin-Dependent Kinase Inhibitor p16; Cyclin-Dependent Kinase Inhibitor p18; 16-fluoroestradiol; Steroids; Hormones; Magnetic Resonance Spectroscopy; High-Energy Shock Waves; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (STEMVAC, ET + CDK4/6i) (Experimental): After completion of 2 cycles of SOC ET + CDK4/6i therapy, patients receive STEMVAC ID on the following schedule: 1) Three "priming" doses every 28 days; 2) Two "booster" doses at 6 and 9 months after "priming" dose #3; and 3) Additional "booster" doses every 6 months in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or ultrasound-guided biopsies, as well as collection of blood samples and CT or PET scans throughout the trial.
  Interventions: Biological: CD105/Yb-1/SOX2/CDH3/MDM2-polyepitope Plasmid DNA Vaccine; Procedure: Computed Tomography; Drug: Cyclin-Dependent Kinase 4 Inhibitor; Drug: Cyclin-Dependent Kinase 6 Inhibitor; Drug: Hormone Therapy; Procedure: Positron Emission Tomography; Procedure: Ultrasound Imaging; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection
- Cohort 2 (STEMVAC, capecitabine) (Experimental): After completion of 1 cycle of SOC capecitabine treatment, patients receive STEMVAC ID on the following schedule: 1) Three "priming" doses every 28 days; 2) Two "booster" doses at 6 and 9 months after "priming" dose #3; and 3) Additional "booster" doses every 6 months in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or ultrasound-guided biopsies, collection of blood samples, and FES PET scans, as well as CT or PET scans throughout the trial.
  Interventions: Biological: CD105/Yb-1/SOX2/CDH3/MDM2-polyepitope Plasmid DNA Vaccine; Drug: Capecitabine; Procedure: Computed Tomography; Drug: F-18 16 Alpha-Fluoroestradiol; Procedure: Positron Emission Tomography; Procedure: Ultrasound Imaging; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection

INTERVENTIONS:
Biological: CD105/Yb-1/SOX2/CDH3/MDM2-polyepitope Plasmid DNA Vaccine — Given ID
  Other Names: STEMVAC; STEMVAC Th1 Polyepitope Plasmid-based Vaccine; CD105/Yb-1/SOX2/CDH3/MDM2 Plasmid Vaccine
Drug: Capecitabine — Given SOC capecitabine
  Other Names: Ro 09-1978/000; Xeloda
  Arms: Cohort 2 (STEMVAC, capecitabine)
Procedure: Computed Tomography — Undergo CT or ultrasound-guided biopsies
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Cyclin-Dependent Kinase 4 Inhibitor — Given SOC CDK4/6i
  Other Names: CDK4 Inhibitor
  Arms: Cohort 1 (STEMVAC, ET + CDK4/6i)
Drug: Cyclin-Dependent Kinase 6 Inhibitor — Given SOC CDK4/6i
  Other Names: CDK6 Inhibitor
  Arms: Cohort 1 (STEMVAC, ET + CDK4/6i)
Drug: F-18 16 Alpha-Fluoroestradiol — Undergo FES PET
  Other Names: 16 alpha-fluroestradiol-17 beta; F-18 FES; FES; Fluorine-18 16 alpha-fluoroestradiol; Fluoroestradiol F-18
  Arms: Cohort 2 (STEMVAC, capecitabine)
Drug: Hormone Therapy — Given SOC ET
  Other Names: Chemotherapy-Hormones/Steroids; Endocrine Therapy; Hormonal; Hormonal Therapy; hormone treatment; Hormones
  Arms: Cohort 1 (STEMVAC, ET + CDK4/6i)
Procedure: Positron Emission Tomography — Undergo PET or FES PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: Ultrasound Imaging — Undergo CT or ultrasound-guided biopsies
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasonography; Ultrasound; Ultrasound Test; Ultrasound, Medical; US
Procedure: Biopsy Procedure — Undergo CT or ultrasound-guided biopsies
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection

SUMMARY:
This phase II trial studies how well a vaccine, STEMVAC, works in combination with standard endocrine-based therapy (ET) with a CDK4/6 targeted drug therapy, or with the chemotherapy drug capecitabine, in treating patients with hormone receptor (HR)-positive, HER2-negative breast cancer that has spread from where it first started (primary site) to other places in the body (metastatic). STEMVAC is designed to target proteins that cancer cells use when they become more aggressive and start to spread, and it is believed to work by boosting the immune system to recognize and destroy the invader tumor cells that are causing the disease. Standard ET is treatment that adds, blocks, or removes hormones in order to slow or stop the growth of cancer. Standard CDK4/6 inhibitors may stop the growth of tumor cells and may kill them by blocking some of the enzymes needed for cell growth. Capecitabine is in a class of medications called antimetabolites. It is taken up by tumor cells and breaks down into fluorouracil, a substance that kills tumor cells. Giving STEMVAC in combination with standard ET or chemotherapy may be an effective treatment for metastatic HR positive, HER2 negative breast cancer.

DETAILED DESCRIPTION:
OUTLINE: Patients with ET-sensitive disease are assigned to Cohort 1, while patients with ET-resistant disease are assigned to Cohort 2.

COHORT 1: After completion of 2 cycles of standard of care (SOC) ET + CDK4/6 inhibitor (CDK4/6i) therapy, patients receive STEMVAC intradermally (ID) on the following schedule: 1) Three "priming" doses every 28 days; 2) Two "booster" doses at 6 and 9 months after "priming" dose #1; and 3) Additional "booster" doses every 6 months in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) or ultrasound-guided biopsies for research purposes, as well as collection of blood samples and CT or positron emission tomography (PET) scans throughout the trial.

COHORT 2: After completion of 1 cycle of SOC capecitabine treatment, patients receive STEMVAC ID on the following schedule: 1) Three "priming" doses every 28 days; 2) Two "booster" doses at 6 and 9 months after "priming" dose #1; and 3) Additional "booster" doses every 6 months in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or ultrasound-guided biopsies for research purposes, collection of blood samples, and fluoroestradiol (FES) positron emission tomography (PET) scans, as well as CT or PET scans throughout the trial.

After completion of study treatment, patients are followed every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least ≥ 18 years of age
* Histologically confirmed hormone receptor positive metastatic breast cancer: Tumors that are positive for estrogen receptor (ER) and/or progesterone receptor (PR)
* HER2-negative or HER2-low will be included and defined as:

  * 0-1+ HER2 expression by immunohistochemistry (IHC) OR
  * Fluorescence in situ hybridization (FISH) negative OR
  * HER2 2+ and FISH negative
  * HER2 low per standard of care in breast cancer
* Patients should be receiving the following therapies to be eligible for the study:

  * Cohort 1: First or second line of endocrine therapy in combination with a CDK4/6 inhibitor. Patients must have completed at least 2 cycles of CDK4/6 inhibitor
  * Cohort 2: Progressed on endocrine-based therapies and after completion of at least 1 cycle of capecitabine
* Subjects with Eastern Cooperative Oncology Group (ECOG) Performance Status Score of 0 or 1
* Metastatic disease that is measurable based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or PET Response Criteria in Solid Tumors (PERCIST). Target lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
* Willing to undergo up to two serial biopsies while on study
* Have at least 1 site of disease confirmed by the treating oncologist that could be biopsied during treatment. Ideally the tumor biopsy should not be a site that is used for RECIST/PERCIST measurement and response to treatment; however, this site may have to be biopsied to adhere to protocol or for patient safety. Lesions that will be biopsied should not be in a previously irradiated area unless progression has been demonstrated in such lesions
* White blood cell (WBC) ≥ 2000/mm^3 (within 28 days of receiving the study vaccine)
* Lymphocyte count ≥ 500/mm^3 (within 28 days of receiving the study vaccine)
* Absolute neutrophil count (ANC) ≥ 800/µL (within 28 days of receiving the study vaccine)
* Platelets ≥ 75,000/µL (within 28 days of receiving the study vaccine)
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN), except patients with Gilbert's syndrome in whom total bilirubin must be ≤ 3.0 mg/dL (within 28 days of receiving the study vaccine)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 3 x institutional upper limit of normal (ULN) (within 28 days of receiving the study vaccine)
* Creatinine ≤ 2.0 mg/dL or creatinine clearance > 30 mL/min (within 28 days of receiving the study vaccine)
* Patients of child-bearing potential must agree to use dual methods of contraception and have a negative urine pregnancy test at screening, and male patients must use an effective barrier method of contraception if sexually active with a female of child-bearing potential. Acceptable methods of contraception are condoms with contraceptive foam, oral, implantable or injectable contraceptives, contraceptive patch, intrauterine device, diaphragm with spermicidal gel, or a sexual partner who is surgically sterilized or postmenopausal. Effective methods of contraception must be used throughout the study and until the end of treatment on study
* Must have recovered from major infections and/or surgical procedures; and in the opinion of the investigator, not have any significant active concurrent medical illnesses or condition precluding protocol treatment

Exclusion Criteria:

* Patients with any of the following cardiac conditions:

  * Symptomatic restrictive cardiomyopathy
  * Dilated cardiomyopathy
  * Unstable angina within 4 months prior to enrollment
  * New York Heart Association functional class III-IV heart failure on active treatment
  * Symptomatic pericardial effusion
  * Uncontrolled hypertension
  * Uncontrolled cardiac arrhythmias
* Patients with any autoimmune disease or comorbidities that require chronic steroids or immunosuppressants
* A non-breast malignancy requiring radiation or systemic therapy within last 5 years
* Known hypersensitivity reaction to the granulocyte-macrophage colony-stimulating factor (GM-CSF) adjuvant; any known contra-indication to GM-CSF
* Pregnant or breast feeding
* Known history of human immunodeficiency virus (HIV) infection, hepatitis B (e.g., hepatitis B virus surface antigen [HBsAg] reactive), or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Major surgery within the 4 weeks prior to initiation of study vaccine
* Current use of immunosuppressive agents or systemic corticosteroids. Topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption) are allowed. Patients who have received systemic corticosteroids ≤ 30 days prior to starting study drug will be excluded
* Patient is currently enrolled in any other clinical protocol or investigational trial that involves administration of experimental therapy and/or therapeutic devices, or investigational drug

  * NOTE: Biomarker or tissue collection or any other non-interventional clinical trial enrollment is allowed
* Must be 14 days between a non-study vaccine and any STEMVAC vaccination

  * NOTE: The minimum of 14 days does not apply to the tetanus and diphtheria (Td) vaccine
* Any condition that may interfere with the patient's participation in the study per treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 3 years after completion of study treatment
  Safety and systemic toxicity will be determined by chemical and clinical parameters evaluated at various time points. Toxicity grading will be evaluated according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 6.0 and monitoring of AEs will be done per Food and Drug Administration and NCI guidelines. The type and grade of toxicities noted during the immunization regimen will be summarized. The duration of toxicities will also be summarized using descriptive statistics such as mean and standard deviation. All AEs noted by the investigator will be tabulated according to the affected body system. The frequency and severity of adverse events will be summarized with a proportion and a 95% confidence interval (CI).
Incidence of immunogenicity | Pre-vaccine up to after 2 booster doses of STEMVAC vaccine (Up to 40 weeks)
  Will be defined as the sum of the interferon gamma enzyme-linked immunosorbent spot of all STEMVAC antigens on blood samples collected pre-vaccine as compared to 1-month post dose #3 of the STEMVAC vaccine and again after 2 booster doses of STEMVAC vaccine. Both incidence and magnitude will be assessed. Immune responses will be summarized with mean and standard deviation or median and range (if skewness is observed) over time, the change over time will be summarized with graphs, and also analyzed using linear mixed-effects regression models with normalizing transformation if necessary.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From the start of treatment to the worsening of cancer as determined by primary treating oncologist or death whichever occurs first, assessed up to 3 years after completion of study treatment
  Will be analyzed using the Kaplan-Meier method. Kaplan-Meier estimates of the survival function with 95% CIs at specific time points (using Greenwood's formula for the standard error) will be computed.
Circulating tumor DNA (ctDNA) | Up to 3 years after completion of study treatment
  Will evaluate persistence and level of ctDNA over time in peripheral blood with addition of STEMVAC at baseline, after completion of priming monthly doses, at booster vaccines, and at progression (end of study). Linear mixed-effects regression models with normalizing transformation (if necessary) will be employed to evaluate changes in ctDNA levels over time. Paired t test or Wilcoxon signed rank tests will be applied for pairwise comparisons (depending on the distribution) between time points.
Elimination of cancer cells associated with epithelial to mesenchymal transformation (EMT) | Up to 3 years after completion of study treatment
  Will determine whether STEMVAC immunization in addition to either endocrine therapy plus a CDK4/6 inhibitor or capecitabine results in elimination of cancer cells associated with EMT, as EMT proteins are targeted by this vaccine. Will determine EMT signature by gene expression profiling in baseline tumor (previously collected tumor biopsy) and compare with post-STEMVAC tumor biopsy. Gene expression profiles from biopsies before and after vaccination will be compared using paired t test or Wilcoxon signed-rank test (depending on the distribution) to determine if vaccination modulates the EMT gene signature in the tumor. Differential gene expression analysis or linear models will be used to analyze individual EMT gene expression levels.

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Hunter, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No